CLINICAL TRIAL: NCT05091411
Title: Randomized, Double-blind, Parallel-controlled Evaluation of the Immunogenicity Consistency and Safety of the Three Batches of Recombinant Novel Coronavirus Vaccine (CHO Cells) After Process Verification in the 18-59-year-old Population, and the Comparison With the Pilot-scale Batch Immunogenicity Non-inferiority Bridging and Safety Clinical Trials
Brief Title: Clinical Trials of the Consistency and Non-inferiority Bridging Between Batches of Recombinant New Coronavirus Vaccine (CHO Cells)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LKM-2021-NCV02
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Coronavirus Disease 2019
Keywords: Recombinant Novel Coronavirus Vaccine
MeSH Terms: conditions — COVID-19 | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Population Ⅰ (Experimental): 3 doses of experimental vaccine (pilot scale batch) were given at day 0, 30 and 60.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell) group
- Population Ⅱ (Experimental): 3 doses of experimental vaccine (process validation lot 1) at day 0, 30 and 60;
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell) group
- Population Ⅲ (Experimental): 3 doses of experimental vaccine (process validation lot 2) at day 0, 30 and 60;
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell) group
- Population Ⅳ (Experimental): 3 doses of experimental vaccine (process validation lot 3) were given at day 0, 30 and 60.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell) group

INTERVENTIONS:
Biological: Recombinant new coronavirus vaccine (CHO cell) group — Intramuscular injection of deltoid muscle of upper arm of 25μg/0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).

SUMMARY:
Popular topic:Clinical trials of the consistency and non-inferiority bridging between batches of recombinant new coronavirus vaccine (CHO cells) Research purpose:Main purpose:1)To evaluate the interbatch consistency of immunogenicity of three batches of recombinant Novel Coronavirus vaccine (CHO cells) following process validation in 18-59 year olds. 2)To evaluate the non-inferiority of immunogenicity of recombinant Novel Coronavirus vaccine (CHO cells) from the combined batch and pilot scale batch after process validation in 18-59 years of age. Secondary purpose:1)To evaluate the safety of each batch of recombinant Novel Coronavirus vaccine (CHO cells) in patients aged 18-59 years.2)To evaluate the non-inferiority of immunogenicity of recombinant Novel Coronavirus vaccine (CHO cells) from the combined batch and commercial batch after process validation in 18-59 years of age.

Overall design:This trial adopts a randomized, double-blind, parallel controlled trial design. Study population:The study involved people aged 18-59. Test groups:A total of 1680 subjects were enrolled in this clinical trial and randomly divided into 4 groups at 1:1:1:1 (pilot scale batch: process verification batch 1: process verification batch 2: process verification batch 3) , 420 cases per group.

DETAILED DESCRIPTION:
Overall design: In this study, a randomized, double-blind, parallel-controlled trial design was used to evaluate the inter-batch consistency of immunogenicity of the three batches of recombinant Novel Coronavirus vaccine (CHO cells) after process validation in 18-59 year olds and the non-inferiority of immunogenicity between the three batches after process validation and the pilot scale batches. Non-inferiority of immunogenicity between the three batches after process validation and the commercial scale batches (clinical trials have been conducted), and the safety of each vaccine batch after vaccination was evaluated.

Intervention: Group A: 3 doses of experimental vaccine (pilot scale batch) were given at day 0, 30 and 60; Group B: 3 doses of experimental vaccine (process validation lot 1) at day 0, 30 and 60; Group C: 3 doses of experimental vaccine (process validation lot 2) at day 0, 30 and 60; Group D: 3 doses of experimental vaccine (process validation lot 3) at day 0, 30 and 60;

Immunogenicity observation:Blood samples were collected before the first dose and 14 days after the whole immunization, and the serum was separated for detection of live virus neutralizing antibodies (CPE method).

Safety observation:

(1) All adverse events (AE) were collected 30 minutes after each dose, all AE (including both solicitation and non-solicitation AE) at 0-7 days, and all AE (non-solicitation AE) at 8-30 days.

Solicitation AE (the following events occurring within 7 days of vaccination) :

1. Adverse events at the inoculation site (local) : pain, swelling, induration, redness, rash, pruritus;
2. Vital signs: fever;
3. Non-inoculated site (systemic) adverse events: headache, fatigue/fatigue, nausea, vomiting, diarrhea, muscle pain (non-inoculated site), cough, acute allergic reactions.

(2) All SAE were collected from the first dose to 12 months after full immunization.

ELIGIBILITY:
Inclusion Criteria:

1. Persons aged 18-59 with full capacity for civil conduct;
2. Subjects voluntarily participate in the study, sign informed consent, provide valid identification, understand and comply with the requirements of the study protocol;
3. Female subjects of reproductive age agree to use effective contraceptive measures from the beginning of the study to 12 months after full vaccination.

Exclusion Criteria:

1. Suspected or confirmed fever within 72 hours before enrollment, or armpit temperature ≥37.3℃ on the day of enrollment;
2. Diastolic blood pressure ≥100mmHg and/or systolic blood pressure ≥160mmHg before screening;
3. people who currently have or have a history of COVID-19;
4. Persons suffering from the following diseases:

   ① have thrombocytopenia, any coagulation dysfunction or receive anticoagulant treatment, etc.;

   ② history of congenital or acquired immune deficiency or autoimmune disease; Received immunomodulators within 6 months, such as immunosuppressive doses of glucocorticoids (dose reference: equivalent to prednisone 20mg/ day, over a week); Or monoclonal antibodies; Or thymosin; Or interferon; However, topical use (such as ointments, eye drops, inhalants or nasal sprays) is allowed;

   ③ Cancer patients (except basal cell carcinoma);

   ④ Patients with active tuberculosis, viral hepatitis and/or HIV antibody positive or syphilis specific antibody positive;

   ⑤ Neurological disease or family history (e.g., migraines, epilepsy, stroke, seizures in the last three years, encephalopathy, focal neurological deficits, Guillain-Barre syndrome, encephalomyelitis or transverse myelitis); History of mental illness or family history;

   ⑥ Functional absence of spleen, and absence of spleen or splenectomy caused by any reason;

   ⑦ Serious chronic diseases or diseases in the advanced stage can not be controlled smoothly, such as diabetes, thyroid diseases;

   ⑧ Severe liver and kidney diseases; Any current respiratory illness requiring routine medication (e.g., chronic obstructive pulmonary disease [COPD], asthma) or any exacerbation of respiratory illness (e.g., exacerbation of asthma) within the last 5 years; A history of serious cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease, arrhythmia, conduction block, myocardial infarction, cor pulmonale) or myocarditis or pericarditis.
5. A history of severe allergy to any vaccine, or to any component of the test vaccine, including aluminum preparations, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, dyspnea, angiopantic edema, etc.;
6. Subunit vaccine and inactivated vaccine should be administered within 14 days before the first dose of vaccine, and live attenuated vaccine should be administered within 30 days;
7. Have received blood or blood-related products, including immunoglobulin, within 3 months; Or planned use from the beginning of the study to 1 month after full vaccination;
8. Those who have participated in or are participating in other CLINICAL trials related to COVID-19, or who have received COVID-19 vaccines;
9. Lactating women or pregnant women (including women of childbearing age with positive urine pregnancy test);
10. The Investigator believes that the subject has any disease or condition that may place the subject at unacceptable risk; Subjects cannot meet the requirements of the program; Conditions that interfere with the assessment of vaccine response.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1680 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity endpoint | 14 days after vaccination
  GMT and positive rate of SARS-COV-2 neutralizing antibody 14 days after vaccination with recombinant Novel Coronavirus vaccine (CHO cells)

CONTACTS AND LOCATIONS:
Overall Officials: Tao Huang, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No